CLINICAL TRIAL: NCT07312851
Title: A Phase I, Randomized, Single-blind, Placebo-controlled Study to Further Characterize Andexanet Posology and Assess the Interaction Between Andexanet and Subsequent Enoxaparin in Healthy Participants
Brief Title: A Study to Investigate Andexanet Dosing and the Interaction Between Andexanet and Subsequent Enoxaparin in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D9609C00001; 2025-522513-30-00 (Other: EUCT Number)
Record Dates: First submitted 2025-11-27; First posted 2025-12-31 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: Posology; Re-anticoagulation; Pharmacodynamics; Life-threatening or uncontrolled bleeding; Thrombotic events; Factor Xa inhibitors
MeSH Terms: interventions — PRT064445; Rivaroxaban; apixaban; Enoxaparin

STUDY DESIGN:
Intervention Model Description: 4 Modules divided into 2 Parts
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Module 1: Rivaroxaban + Andexanet (dose A) (Experimental): Participants will receive once daily dose of 20 mg rivaroxaban from Day -3 to Day -1 to achieve steady state plasma levels. On Day 1, approximately 3 hours before andexanet (dose A) dosing, the participants will receive an additional dose of rivaroxaban. Participants will be further allocated to groups to receive doses of enoxaparin at different time points after the end of andexanet bolus.
  Interventions: Drug: Andexanet alfa; Drug: Rivaroxaban; Drug: Enoxaparin
- Module 1: Rivaroxaban + Andexanet (dose B) (Experimental): Participants will receive once daily dose of 20 mg rivaroxaban from Day -3 to Day -1 to achieve steady state plasma levels. On Day 1, approximately 3 hours before andexanet (dose B) dosing, the participants will receive an additional dose of rivaroxaban.
  Interventions: Drug: Andexanet alfa; Drug: Rivaroxaban
- Module 1: Rivaroxaban + Andexanet (dose C) (Experimental): Participants will receive once daily dose of 20 mg rivaroxaban from Day -3 to Day -1 to achieve steady state plasma levels. On Day 1, approximately 3 hours before andexanet (dose C) dosing, the participants will receive an additional dose of rivaroxaban.
  Interventions: Drug: Andexanet alfa; Drug: Rivaroxaban
- Module 1: Rivaroxaban + Placebo (Experimental): Participants will receive once daily dose of 20 mg rivaroxaban from Day -3 to Day -1 to achieve steady state plasma levels. On Day 1, approximately 3 hours before placebo (equivalent to dose B of andexanet) dosing, the participants will receive an additional dose of rivaroxaban. Participants will be further allocated to groups to receive doses of enoxaparin at different time points after placebo administration.
  Interventions: Drug: Rivaroxaban; Drug: Enoxaparin; Other: Placebo
- Module 2: Apixaban + Andexanet (dose B) (Experimental): Participants will receive twice daily dose of 5 mg apixaban from Day -3 to Day -1 to achieve steady state plasma levels. On Day 1, approximately 3 hours before andexanet (dose B) dosing, the participants will receive an additional dose of apixaban. Participants will be further allocated to groups to receive doses of enoxaparin at different time points after the end of andexanet bolus.
  Interventions: Drug: Andexanet alfa; Drug: Apixaban; Drug: Enoxaparin
- Module 2: Apixaban + Andexanet (dose C) (Experimental): Participants will receive twice daily dose of 5 mg apixaban from Day -3 to Day -1 to achieve steady state plasma levels. On Day 1, approximately 3 hours before andexanet (dose C) dosing, the participants will receive an additional dose of apixaban.
  Interventions: Drug: Andexanet alfa; Drug: Apixaban
- Module 2: Apixaban + Andexanet (dose D) (Experimental): Participants will receive twice daily dose of 5 mg apixaban from Day -3 to Day -1 to achieve steady state plasma levels. On Day 1, approximately 3 hours before andexanet (dose D) dosing, the participants will receive an additional dose of apixaban.
  Interventions: Drug: Andexanet alfa; Drug: Apixaban
- Module 2: Apixaban + Placebo (Experimental): Participants will receive twice daily dose of 5 mg apixaban from Day -3 to Day -1 to achieve steady state plasma levels. On Day 1, approximately 3 hours before placebo (equivalent to dose B of andexanet) dosing, the participants will receive an additional dose of apixaban. Participants will be further allocated to groups to receive doses of enoxaparin at different time points after placebo administration.
  Interventions: Drug: Apixaban; Drug: Enoxaparin; Other: Placebo
- Module 3: Rivaroxaban + Andexanet (Dose A) (Experimental): Participants will receive once daily dose of 20 mg rivaroxaban from Day -3 to Day -1 to achieve steady state plasma levels. On Day 1, approximately 3 hours before andexanet (dose A) dosing, the participants will receive an additional dose of rivaroxaban.
  Interventions: Drug: Andexanet alfa; Drug: Rivaroxaban
- Module 3: Apixaban + Andexanet (Dose B) (Experimental): Participants will receive twice daily dose of 5 mg apixaban from Day -3 to Day -1 to achieve steady state plasma levels. On Day 1, approximately 3 hours before andexanet (dose B) dosing, the participants will receive an additional dose of apixaban.
  Interventions: Drug: Andexanet alfa; Drug: Apixaban
- Module 3: Rivaroxaban + Placebo (Experimental): Participants will receive once daily dose of 20 mg rivaroxaban from Day -3 to Day -1 to achieve steady state plasma levels. On Day 1, approximately 3 hours before placebo (equivalent to dose A of andexanet) dosing, the participants will receive an additional dose of rivaroxaban.
  Interventions: Drug: Rivaroxaban; Other: Placebo
- Module 3: Apixaban + Placebo (Experimental): Participants will receive twice daily dose of 5 mg apixaban from Day -3 to Day -1 to achieve steady state plasma levels. On Day 1, approximately 3 hours before placebo (equivalent to dose B of andexanet) dosing, the participants will receive an additional dose of apixaban.
  Interventions: Drug: Apixaban; Other: Placebo
- Module 4: Placebo + Andexanet (dose C) (Experimental): Participants will receive daily dose of one placebo tablet from Day -3 to Day -1. On Day 1, approximately 3 hours before andexanet (dose C) dosing, the participants will receive an additional placebo tablet.
  Interventions: Drug: Andexanet alfa; Other: Placebo
- Module 4: Placebo + Andexanet (dose B) (Experimental): Participants will receive daily dose of one placebo tablet from Day -3 to Day -1. On Day 1, approximately 3 hours before andexanet (dose B) dosing, the participants will receive an additional placebo tablet. Participants will be further allocated to groups to receive doses of enoxaparin at different time points after the end of andexanet bolus.
  Interventions: Drug: Andexanet alfa; Drug: Enoxaparin; Other: Placebo

INTERVENTIONS:
Drug: Andexanet alfa — Andexanet alfa will be administered as an intravenous bolus followed by an infusion, however, in Module 3, only a bolus will be given.
  Arms: Module 1: Rivaroxaban + Andexanet (dose A); Module 1: Rivaroxaban + Andexanet (dose B); Module 1: Rivaroxaban + Andexanet (dose C); Module 2: Apixaban + Andexanet (dose B); Module 2: Apixaban + Andexanet (dose C); Module 2: Apixaban + Andexanet (dose D); Module 3: Apixaban + Andexanet (Dose B); Module 3: Rivaroxaban + Andexanet (Dose A); Module 4: Placebo + Andexanet (dose B); Module 4: Placebo + Andexanet (dose C)
Drug: Rivaroxaban — Rivaroxaban will be administered as an oral tablet.
  Arms: Module 1: Rivaroxaban + Andexanet (dose A); Module 1: Rivaroxaban + Andexanet (dose B); Module 1: Rivaroxaban + Andexanet (dose C); Module 1: Rivaroxaban + Placebo; Module 3: Rivaroxaban + Andexanet (Dose A); Module 3: Rivaroxaban + Placebo
Drug: Apixaban — Apixaban will be administered as an oral tablet.
  Arms: Module 2: Apixaban + Andexanet (dose B); Module 2: Apixaban + Andexanet (dose C); Module 2: Apixaban + Andexanet (dose D); Module 2: Apixaban + Placebo; Module 3: Apixaban + Andexanet (Dose B); Module 3: Apixaban + Placebo
Drug: Enoxaparin — Enoxaparin will be administered as a subcutaneous injection.
  Arms: Module 1: Rivaroxaban + Andexanet (dose A); Module 1: Rivaroxaban + Placebo; Module 2: Apixaban + Andexanet (dose B); Module 2: Apixaban + Placebo; Module 4: Placebo + Andexanet (dose B)
Other: Placebo — Placebo will replace andexanet and be given as an IV bolus plus infusion in Modules 1 and 2; in Module 3, placebo will be IV bolus only. In Module 4, an oral placebo tablet will replace rivaroxaban and apixaban.
  Arms: Module 1: Rivaroxaban + Placebo; Module 2: Apixaban + Placebo; Module 3: Apixaban + Placebo; Module 3: Rivaroxaban + Placebo; Module 4: Placebo + Andexanet (dose B); Module 4: Placebo + Andexanet (dose C)

SUMMARY:
The purpose of this study is to characterize andexanet posology and interaction between andexanet and enoxaparin post infusion in healthy participants.

DETAILED DESCRIPTION:
This is a single-blind, placebo-controlled study. The study has 4 modules, which is then divided into 2 parts. Part A of the study will focus on further characterization of andexanet posology and Part B of the study will evaluate a re-institution of anticoagulation with enoxaparin.

Module 1, 2 and 4 - rivaroxaban, apixaban and enoxaparin: These modules are designed to determine the pharmacodynamic (PD) effect of andexanet by assessing its reversal effects on rivaroxaban and apixaban anticoagulation, or assessing its effects in the absence of anticoagulants, and to identify the time interval after andexanet administration at which andexanet shows no impact on enoxaparin.

Module 3 - rivaroxaban and apixaban: This Module is designed to determine the PD effect of bolus only andexanet by assessing its reversal effect on rivaroxaban and apixaban anticoagulation.

All the Modules will comprise:

* A Screening/Enrollment Period of maximum 28 days.
* An in-house stay comprising of a safety baseline lab period (Day -3 to Day -1)
* Treatment period (Day 1 to Day 2)
* Safety follow-up period (Day 3 to Day 5)
* A final Follow-up Visit within 30 days (+7 days) after the last andexanet/placebo administration.

ELIGIBILITY:
Main Inclusion Criteria:

* All females must have a negative pregnancy test at the Screening Visit.
* Females of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the study specific contraception methods.
* Have a Body Mass Index (BMI) between 18.5 and 30.0 kg/m2 (both inclusive) and weigh at least 60 kg.
* Agree to abstain from alcohol consumption or smoking for the duration of the residential period, and from the use of drugs of abuse for the duration of the study.
* Be in good health and agree to have any dietary or nutritional supplements, if needed.

Main Exclusion Criteria:

* History of any clinically significant disease or disorder which may either put the participant at risk because of participation in the study or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of abnormal bleeding or bleeding disorders (eg, hemophilia, von Willebrand disease), signs or symptoms of active bleeding, or risk factors for bleeding.
* History of adult asthma or chronic obstructive pulmonary disease or current regular or as needed use of inhaled medications.
* Family history of or known risk factors for a hypercoagulable or thrombotic condition or thrombotic event, such as anti-phospholipid syndrome; Factor V Leiden carrier or homozygote; Protein C, S, or AT3 activity below the normal range.
* Past or current medical history of thrombosis, any sign or symptom that suggests an increased risk of a systemic thrombotic condition, or recent events that may increase risk of thrombosis.
* Any medical or surgical conditions which may impair drug (anticoagulant or andexanet) uptake, metabolism, or excretion.
* An absolute or relative contraindication to anticoagulation or treatment with apixaban, rivaroxaban or enoxaparin.
* Any clinically significant illness or medical procedure within 4 weeks of the first administration of study intervention.
* Any clinically significant abnormalities in clinical chemistry, hematology, coagulation or urinalysis results
* Any positive result on Screening for serum hepatitis B surface antigen (HBsAg) OR anti-hepatitis B core (HBc) antibody, indicative of active hepatitis B (ie, participants with positive anti-HBc antibody result are acceptable if anti-HBc IgM antibodies are negative), anti- hepatitis C virus (HCV) or human immunodeficiency virus (HIV).
* History of severe allergy/hypersensitivity or ongoing clinically significant allergy/hypersensitivity, including heparin-induced thrombocytopenia, or history of hypersensitivity to drugs with a similar chemical structure or class to andexanet, apixaban, rivaroxaban, or enoxaparin or any of the vehicle ingredients.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, intake of > 3 × daily recommended levels of vitamins and minerals during the 2 weeks prior to the first administration of study intervention or longer (> 5 half-lives) if the medication has a long half-life. The participant has taken (by any route) one or more doses of aspirin (including baby aspirin), salicylate or subsalicylate, other antiplatelet drugs (eg, ticagrelor, clopidogrel, ticlopidine), non-steroidal anti-inflammatory drugs, fibrinolytic, or any anticoagulant within 7 days prior to Admission or is anticipated to require such drugs during the study. The participant has been receiving (by any route) hormonal contraception, postmenopausal HRT (including over-the-counter products), or testosterone during the 4 weeks prior to Admission or is anticipated to require such drugs during the study.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days or 5 half-lives (whichever is longest) of Admission.
* Participants who have previously received andexanet.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 186 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Anti-Factor (F) Xa activity | Day 1 post dose
  To determine the pharmacodynamic (PD) effect of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation measured by chromogenic enzymatic anti-FXa activity assays.
Change from baseline in anti-FXa activity | Day 1 post dose
  To determine the PD effect of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation measured by chromogenic enzymatic anti-FXa activity assays.
Thrombin generation potential | Day 1 post dose
  To determine the PD effect of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation measured as thrombin generation potential (including Endogenous Thrombin Potential [ETP]).
Change from pre-direct oral anticoagulants (DOAC) in thrombin generation potential | Day 1 post dose
  To determine the PD effect of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation measured as thrombin generation potential (including ETP).
Change from baseline in thrombin generation potential | Day 1 post dose
  To determine the PD effect of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation measured as thrombin generation potential (including ETP).
Time to onset of coagulation | Day 1 post dose
  To determine the PD effect of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation measured as time to onset of coagulation.
Change from pre-DOAC in time to onset of coagulation | Day 1 post dose
  To determine the PD effect of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation measured as time to onset of coagulation.
Change from baseline in time to onset of coagulation | Day 1 post dose
  To determine the PD effect of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation measured as time to onset of coagulation.
Anti-FXa activity following enoxaparin dosing | From Day 1 to Day 2
  To determine anticoagulation by enoxaparin at different time points after andexanet treatment measured by chromogenic enzymatic anti-FXa activity assays.
Thrombin generation potential following enoxaparin dosing | From Day 1 to Day 2
  To determine anticoagulation by enoxaparin at different time points after andexanet treatment measured as thrombin generation potential (including ETP).

SECONDARY OUTCOMES:
Module 3: Anti-FXa activity | Day 1 post dose
  To describe the PD effect of andexanet bolus by assessing reversal of rivaroxaban or apixaban anticoagulation, as measured by chromogenic enzymatic anti-FXa activity assays.
Module 3: Change from baseline in anti-FXa activity | Day 1 post dose
  To describe the PD effect of andexanet bolus by assessing reversal of rivaroxaban or apixaban anticoagulation, as measured by chromogenic enzymatic anti-FXa activity assays.
Module 3: Thrombin generation potential | Day 1 post dose
  To describe the PD effect of andexanet bolus by assessing reversal of rivaroxaban or apixaban anticoagulation, as measured by thrombin generation potential (including ETP).
Module 3: Change from baseline in thrombin generation potential | Day 1 post dose
  To describe the PD effect of andexanet bolus by assessing reversal of rivaroxaban or apixaban anticoagulation, as measured by thrombin generation potential (including ETP).
Module 3: Change from pre-DOAC in thrombin generation potential | Day 1 post dose
  To describe the PD effect of andexanet bolus by assessing reversal of rivaroxaban or apixaban anticoagulation, as measured by thrombin generation potential (including ETP).
Module 3: Time to onset of coagulation | Day 1 post dose
  To describe the PD effect of andexanet bolus by assessing reversal of rivaroxaban or apixaban anticoagulation, as measured by time to onset of coagulation.
Module 3: Change from pre-DOAC in time to onset of coagulation | Day 1 post dose
  To describe the PD effect of andexanet bolus by assessing reversal of rivaroxaban or apixaban anticoagulation, as measured by time to onset of coagulation.
Module 3: Change from baseline in time to onset of coagulation | Day 1 post dose
  To describe the PD effect of andexanet bolus by assessing reversal of rivaroxaban or apixaban anticoagulation, as measured by time to onset of coagulation.
Tissue factor pathway inhibitor (TFPI) activity | Up to Day 4
  To describe additional PD effects of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation on levels of TFPI activity measured by enzymatic TFPI activity assay.
Antithrombin 3 (AT3) | Up to Day 4
  To describe additional PD effects of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation on levels of AT3 measured by an AT3 enzyme-linked immunosorbent assay (ELISA).
Thrombinantithrombin complex (TAT) | Up to Day 4
  To describe additional PD effects of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation on levels of TAT.
Fibrin degradation fragment (D-dimer) | Up to Day 4
  To describe additional PD effects of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation on levels of D-dimer.
Prothrombin fragment 1+2 (F1+2) | Up to Day 4
  To describe additional PD effects of andexanet doses by assessing reversal of rivaroxaban or apixaban anticoagulation on levels of F1+2.

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Berlin, Germany
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/